CLINICAL TRIAL: NCT04374552
Title: RCT in Asymptomatic Volunteers With COVID-19 Comparing Azithromycin and Hydroxychloroquine vs. Hydroxychloroquine Alone vs Standard of Care Without Antibiotics
Brief Title: Asymptomatic COVID-19 Trial
Acronym: ACT
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The investigators have decided not to go forward with this protocol
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Jeffrey L Carson, MD, Distinguished Professor of Medicine, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro2020000872
Record Dates: First submitted 2020-05-02; First posted 2020-05-05 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-05

CONDITIONS: SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine; Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study medication will be tablets containing either active drug or placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Hydroxychloroquine & Azithromycin (Experimental): Hydroxychloroquine sulfate 400 mg po BID for day one and then 400 mg QD for 4 days Azithromycin 500 mg po on day one, followed by 250 mg po QD X 4 days
  Interventions: Drug: Hydroxychloroquine sulfate &Azithromycin
- Placebo (Placebo Comparator): Placebo for Hydroxychloroquine sulfate (2 pills bid day one and then 2 tablets QD for 4 days) Placebo for Azithromycin (2 pills on day one and followed by 1 pill po QD x 4 days)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydroxychloroquine sulfate &Azithromycin — Drug - Hydroxychloroquine sulfate &Azithromycin
  Arms: Hydroxychloroquine & Azithromycin
Drug: Placebo — Drug - placebo
  Arms: Placebo

SUMMARY:
The coronavirus disease-2019 (COVID-19) is spreading throughout the United States. While there are no known therapies to treat those who have become sick, there have been some reports that a medication currently used to treat rheumatoid arthritis, lupus, and malaria (Hydroxychloroquine sulfate, also known as Plaquenil) may help to lessen the chance or severity of illness, especially if combined with a medicine that treats other kinds of infections (Azithromycin, also known as Zithromax or Zmax or Zpak).

There are some people who test positive for the virus but who are otherwise not ill. Current standard of care is to advise these people to self-monitor but no treatment is offered. It is not known how many of these individuals will remain symptom free, and how many will become sick or how severe those symptoms will be. This study will randomize those people who do not have symptoms into one of three treatment plans 1) Hydroxycholoquine and Azithromycin, or 2) no active medication (placebo). All participants will be followed for 2 months.

The study will determine if there is any benefit to those who are asymptomatic to taking taking Hydroxychloroquine sulfate in combination with Azithromycin, or if there is no benefit from taking these medications.

DETAILED DESCRIPTION:
Participants will be randomized into one of two treatment plans

1. Hydroxycholoquine sulfate in combination with Azithromycin Hydroxycholorquine as above, plus Azithromycine: 500 mg po for day 1and then 250 mg QD for 4 days
2. no active medication (placebo)

All participants will be followed for 2 months. The primary aim is to determine if there is any benefit (reduced likelihood for development of fever and other symptoms of COVID-19 ) to taking only Hydroxychloroquine sulfate, or to taking Hydroxychloroquine sulfate in combination with Azithromycin, or if there is no benefit to taking these medications for this population.

ELIGIBILITY:
Inclusion Criteria:

1. Documented SARS-CoV-2 infection by qPCR assay without symptoms consistent with COVID-19 within 1 week of enrollment
2. Age ≥20

Exclusion Criteria:

1. Retinal eye disease
2. Known glucose-6 phosphate dehydrogenase (G-6-PD) deficiency
3. Known chronic kidney disease, stage 4 or 5 or receiving dialysis
4. Current use of:

   * Class 3 AAD - amiodarone, dronaderone, dofetilide, sotalol)
   * Class 1A AAD (procainamide, quinidine, disopyramide)
   * Flecainide
   * chlorpromazine
   * Cilostazol (Pletal)
   * Donepezil (Aricept)
   * Droperidol
   * Fluconazole
   * Methadone
   * Ondansetron(Zofran)
   * Thioridazine
   * Macrolides (clarithromycin, erythromycin)
   * Fluroquinolones (ciprofloxacin, levofloxacin, moxifloxacin)
5. Pregnancy or women who are breast feeding
6. Inability to tolerate oral medications
7. Allergy or prior adverse reaction to either azithromycin or hydroxychloroquine sulfate
8. Allergy to adhesives
9. QTc interval > 450 mSEC for men and women
10. History of Torsade de Pointes VT or prior cardiac arrest or congenital long QT interval
11. Non-English-speaking

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-05 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is the rate of decline in viral load over the 10 days after randomization | 10 days
  Change in SARS-CoV-2 viral from baseline to day 6

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Carson, MD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Robert Wood Johnson University Hospital, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided